CLINICAL TRIAL: NCT02154997
Title: The Effect of Different Food Products on Post Prandial Blood Glucose in Pregnant Woman With Diabetes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Uri Elchalal (Other)
Responsible Party: Sponsor-Investigator, Uri Elchalal, Associate Professor Obstetrics and Gynecology Dept, Hadassah Medical Organization
Organization: Hadassah Medical Organization (Other)
Other Study IDs: HMO-0071-14
Record Dates: First submitted 2014-06-02; First posted 2014-06-04 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes; Gestational Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes, Gestational

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Type 1 and Type 2 Diabetes: pregnant women which have a known condition of type 1 or type 2 diabetes
- Gestational diabetes: pregnant women which have developed Gestational diabetes
- Control group: Pregnant women whom do not suffer from any altered glucose metabolism

SUMMARY:
During pregnancy nutrition demands change and the pregnant woman needs to adjust her food intake and take into consideration the corrected daily recommendations for micro and macro nutrients. Pregnant woman tend to suffer from hyperemesis and this affects their food choice.

Amongst pregnant women with Diabetes the glucose balance is extremely important during pregnancy. Glucose balance is a result of correct nutrition and an exact amount of insulin. This delicate balance requires from the pregnant women an ability to perform correct carbohydrate count.

Hyperglycemia has already been proven to affect the fetus and the neonatal outcomes. Hypoglycemia may also have a negative effect but the main danger is immediate harm to the mother and therefore to the fetus. For those reasons glucose balance is crucial and demands delicate synchronization of nutrition and insulin therapy.

ELIGIBILITY:
Inclusion Criteria:

* age 18-45
* women who suffer from type 1 diabetes, type 2 diabetes or gestational diabetes
* Do not suffer from any intestinal disease
* Accept to sign a consent form

Exclusion Criteria:

* over age of 45
* under age of 18
* suffer from any intestinal disease
* do not accept to sign a consent form

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women perticapting in this study will be from the high risk pregnancy clinic of hadassah Ein Kerem.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-11; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Post prandial blood glucose levels | The outcome will be measured at various time points during a 120 min OGTT: Fasting, 30, 60, 90 and 120 min
  For every time point blood glucose will be analyzed for blood glucose and for Insulin and C-peptide for the control group

CONTACTS AND LOCATIONS:
Overall Officials: Ram Weiss, Md PhD, Principal Investigator — Hebrew Universtity; Karen J Hershkop, PhD, Principal Investigator — Hebrew University; Limor Marko, MSc, Principal Investigator — Hebrew University
Locations (1):
- Hadassah Ein Kerem, Jerusalem, Israel